CLINICAL TRIAL: NCT05496062
Title: Evaluation of the Toffee Nasal and Toffee Nasal Pillows Mask in Home, USA, 2022
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIA-305
Record Dates: First submitted 2022-08-08; First posted 2022-08-10 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Obstructive Sleep Apnea
Keywords: Positive Airway Pressure Therapy
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- F&P Toffee Nasal and Toffee Nasal Pillows Mask (Experimental): Participants will be placed in the experimental arm for 14 days, during which they will be using either the Toffee Nasal or Toffee Nasal Pillows mask for PAP therapy.
  Interventions: Device: F&P Toffee Nasal and Toffee Nasal Pillows Masks

INTERVENTIONS:
Device: F&P Toffee Nasal and Toffee Nasal Pillows Masks — F&P Toffee Nasal and Toffee Nasal Pillows Masks are intended to be used within the traditional PAP therapy system and are designed to facilitate equivalent PAP therapeutic efficacy as defined by standard practice.

SUMMARY:
This clinical investigation is designed to assess the F&P Toffee Nasal and Toffee Nasal Pillows masks in home for use during PAP therapy delivery.

The objectives of the investigation are to assess therapeutic efficacy, safety and comfort.

DETAILED DESCRIPTION:
This clinical investigation is designed to assess the F&P Toffee Nasal and Toffee Nasal Pillows masks in home for use during PAP therapy delivery. A target recruitment goal of 45, current PAP therapy users per mask type (e.g. Nasal and Nasal Pillows) will be recruited to participate in this investigation to achieve a total sample of 90. The investigation will involve participation in a two week in home trial of the F&P Toffee Nasal or Toffee Nasal Pillows mask.

The objectives of the investigation are to assess therapeutic efficacy, safety and comfort.

ELIGIBILITY:
Inclusion Criteria:

1. Persons who are ≥ 22 years of age
2. Persons who weigh ≥ 66 lbs (30 kgs)
3. Persons who have been prescribed PAP (APAP, BPAP or CPAP) therapy by a physician
4. Persons who are compliant with PAP therapy for ≥ 4 hours per night for 70% of nights for at least two weeks prior to enrolment in the trial
5. Persons who are currently using either a nasal, sub-nasal or nasal pillows mask
6. Persons who have an IPAP pressure of < 20 cmH2O
7. Persons who currently use a PAP therapy device with data recording capabilities
8. Persons who are fluent in spoken and written English
9. Persons who possess the capacity to provide informed consent

Exclusion Criteria:

1. Persons who are intolerant to PAP therapy
2. Persons who are required to use PAP therapy for more than 12 hours per day or for extensive periods other than sleep or naps
3. Persons using full face masks
4. Persons who possess, or suffer from, anatomical or physiological conditions which make PAP therapy inappropriate
5. Persons who are pregnant or think they may be pregnant
6. Persons who use a PAP therapy machine for the delivery of medicines, except supplemental O2

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2022-09-12 (Actual); Primary Completion 2022-10-07 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Therapeutic Efficacy | After two weeks of use
  The F&P Toffee Nasal and Toffee Nasal Pillows masks provides adequate PAP therapy when used in a home environment. This is an objective measure and is determined by the Apnea-Hypopnea Index recorded on PAP therapy machines after 14 days of use.

SECONDARY OUTCOMES:
Comfort | After two weeks of use
  The F&P Toffee Nasal and Toffee Nasal Pillows is comfortable during PAP therapy when used in a home environment. This is a subjective measure and is determined by a five-point Likert-type scale as recorded on a questionnaire after 14 days of use.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Clinical Site Partners, LLC - DBA CSP Miami, Miami, Florida
  - Clayton Sleep Institute, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: Undecided